CLINICAL TRIAL: NCT06453668
Title: A 52-week, Phase 1 Safety, Pharmacokinetic and Pharmacodynamic Trial of Siplizumab in Newly Diagnosed Adult Amyotrophic Lateral Sclerosis (ALS) Patients (AURORA)
Brief Title: A Study of TCD601 (Siplizumab) in Newly Diagnosed Adult Amyotrophic Lateral Sclerosis (ALS) Patients
Acronym: AURORA
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ITB-Med LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TCD601H101
Record Dates: First submitted 2024-05-06; First posted 2024-06-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-09

CONDITIONS: ALS
Keywords: Amyotrophic Lateral Sclerosis; Neuroinflammatory
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — siplizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): TCD601 (siplizumab) administered with the contemporary standard of care regimen.
  Interventions: Biological: TCD601

INTERVENTIONS:
Biological: TCD601 — Investigational Product
  Other Names: siplizumab

SUMMARY:
The purpose of this study is to investigate the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of TCD601 (siplizumab) in newly diagnosed adult ALS patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female patients ≥ 18 to 80 years of age.
* Diagnosis of ALS by revised El Escorial Criteria, at study entry within 24 months of first symptoms.
* Patients on existing ALS treatment must have been on a stable dose for 28 days.

Key Exclusion Criteria:

* Patient with severe systemic infections, current or within the two weeks prior to randomization.
* Subjects who, in the opinion of the investigator, are not capable of giving informed consent for the study or who are unable or unwilling to adhere to the study requirements outlined in the protocol.
* Use of other investigational products or treatment in another investigational drug study within 30 days of screening
* Pregnant or nursing (lactating) women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the safety of TCD601 in adult patients with ALS | 12 Months
  Assess the incidence of treatment-emergent Adverse Events [Safety and Tolerability]

SECONDARY OUTCOMES:
Evaluation of the pharmacokinetics (PK) | 12 Months
  Siplizumab concentration over time
Correlation of ALS disease status with leucocyte phenotypic profiles | 12 Months
Evaluation of levels of biomarkers | 12 Months
  Neurofilament light chain levels over time
Length of time from trial entry to tracheostomy / death | 12 Months
Assessment of clinically relevant changes in laboratory measurements | 12 Months
  Incidence of abnormal laboratory values
Evaluation of pharmacodynamics (PD) of TCD601 | 12 Months
  Lymphocyte counts by subset over time
Assessment of clinically relevant changes in vital signs | 12 Months
  Incidence of abnormal vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Julin, Study Director — ITB-Med LLC
Locations (3):
- Sweden (3):
  - Skåne University Hospital Malmö, Malmo
  - Studieenheten Akademiskt Specialistcentrum, Stockholm
  - Umeå University Hospital, Umeå